CLINICAL TRIAL: NCT06383481
Title: The Effect of Mobile-Based Education on Postoperative Recovery and Quality of Life in Thyroidectomy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Beyzanur Kızıloğlu, phd student, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TDK-2024-13362
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Diseases; Healthy Lifestyle; Thyroid
Keywords: Thyroidectomy; Patient; Mobile-Based Education; Postoperative Recovery; Quality of Life
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): After the mobile application is introduced to the patients, "T-CSUQ-SV" will be applied first. Following the introduction and information of the mobile application, the "Introductory Information Form, GKAÖ, BARÖ, VHI-10, SF-36 Quality of Life Scale" will be filled out face to face with the patients 1 day before the surgery. The mobile application will be available to the patient. On the first day after the surgery, patients will fill out the GKAÖ, VHI-10, Postoperative Recovery Index, and SF-36 Quality of Life Scale. During each meeting with patients, reminders will be given for the use of the mobile application, and it will be recommended that they read the information in the education section of the mobile application. In the 1st week after the surgery, patients will fill out GKAÖ, BARÖ, VHI-10, and Postoperative Recovery Index. At the 4th and 12th weeks after the surgery, patients will fill out the GKAÖ, BARÖ, VHI-10, Postoperative Recovery Index, SF-36 Quality of Life Scale.
  Interventions: Other: Mobile based education
- Control Group (No Intervention): Control Group Patients in the control group will be provided with standard patient care and information. No application will be made. In summary, week 1 data collection forms will be filled out with the patients at the end of the first week. At the end of the 1st month, 1st month data collection forms will be filled out. At the end of the 3rd month, the study will be terminated by filling out the 3rd month data collection forms.

INTERVENTIONS:
Other: Mobile based education — Control Group Patients in the control group will be provided with standard patient care and information. No application will be made.
  Experimental group The mobile application will be downloaded to the phones of patients who can use the mobile application. The mobile application will be available to the patient. Patients will be informed about daily monitoring of the mobile application, following the training steps, and that they can reach the researcher with consultancy services whenever they need. The mobile application will be made available to patients within a 12-week period and patient follow-up will be provided.
  Arms: Experimental group

SUMMARY:
Thyroid diseases constitute one of the most common health problems around the world and in our country. In its treatment; Drug therapy, radioactive iodine therapy and surgical treatment can be applied alone or together. Advances in the diagnosis of thyroid diseases have led to an increase in the number of thyroidectomies. When there are no complications after thyroidectomy, patients are discharged from the hospital on the day of surgery or are hospitalized for only a few days. In this context, since technical care is given priority, discharge training remains incomplete.

Patients who have had thyroidectomy are discharged within 1-2 days after surgery if no problems occur. For this reason, patient education provided by health professionals and especially nurses may be insufficient. Post-discharge patient education in surgical services can sometimes be ignored, and it is noteworthy that this situation is not given importance due to the busy nature of surgical services. Although short hospital stays after surgery are beneficial in many ways, it increases the need for patient education.

In this study, a mobile application that covers the entire perioperative process and includes education will be developed for patients undergoing thyroidectomy. This developed mobile application aims to manage post-operative problems such as neck pain and discomfort and voice changes experienced by patients, and to improve post-operative recovery, voice quality and, accordingly, quality of life. In this context, it is believed that even in cases where patients cannot access health care professionals, their educational needs will be met, problem management will be provided with applications for the problems they experience, and accordingly, their post-operative recovery, voice and quality of life will increase, starting from the hospital before the surgery until the end of the recovery period, including the home care process after discharge.When the literature on the subject is examined, studies involving education in patients with thyroidectomy are limited. However, no studies have been found on mobile health applications that include training to reduce neck pain and discomfort experienced by thyroidectomy patients, ensure postoperative recovery, and improve voice quality and quality of life.

DETAILED DESCRIPTION:
Thyroid diseases constitute one of the common health problems around the world. In treatment according to the patient's condition; Drug treatment, radioactive iodine treatment and surgical treatment can be applied alone or together. Thyroid surgery; Although its morbidity and mortality rates are low, it is one of the risky and very important surgeries for patients due to the anatomical location and function of the thyroid and the life-threatening complications that may occur. The purpose of thyroid surgery is; It is to complete the surgery with the lowest complications without negatively affecting the success of the surgery and the quality of life. Preoperative patient preparation and meticulous postoperative nursing care are required to prevent complications that may occur during and after thyroidectomy. Focus of post-thyroidectomy care; It is to minimize, prevent or early identify complications and problems that may develop specific to the surgery. When complications do not occur after thyroidectomy, patients are discharged from the hospital on the day of surgery or are hospitalized for only a few days.

It is observed that there are shortenings in hospital stay with the use of ERAS Protocols in patient care. Although short hospital stays are beneficial in many respects, they prevent the patient and family from communicating with health care professionals, shorten the duration of nurse-patient communication and interaction, and increase the need for education and counseling. The ERAS protocol directs surgical nurses to patient education due to the short duration of hospital stay. For this reason, nurses prioritize technical care and discharge training remains inadequate. Having surgery is an important situation in every person's life. Patients need to receive information about the surgery period. It has been shown in the literature that patients' learning needs after thyroidectomy are high and the majority of patients do not have sufficient knowledge. A study found that the implementation of evidence-based nursing guidelines for thyroidectomy patients improved health outcomes and reduced the overall postoperative complication rate by significantly increasing patients' knowledge, practice, and compliance with discharge recommendations. Therefore, patient education after thyroidectomy; It should address the need for information about the surgical procedure, expected postoperative symptoms, wound care, monitoring prescribed medication use, head and neck stretching exercises to reduce neck pain and disability, improving voice quality, monitoring signs of complications, and scheduling follow-up appointments. The information given by the nurse during the surgery positively affects the patient's health outcomes. In order to increase patient comfort and satisfaction, it is very important to implement the education that begins before the surgery and continues until discharge, supported by different educational materials. With developing technology, written materials have been replaced by online platforms. Web-based training provided by nurses strengthens the patient-nurse relationship and draws attention to the educational role of nurses, who play a key role in the preoperative period.

As in patients after all surgical interventions, various postoperative physical, social, mental and functional problems may be observed in patients with thyroidectomy. Patients who undergo thyroid surgery often experience uncomfortable problems such as neck pain, shoulder stiffness, difficulty in shoulder movements, suffocation, feeling of pressure or discomfort, and hoarseness. These problems can continue for a long time after surgery and affect the daily life of patients in a holistic way. Such symptoms are often transient but can still negatively impact both disease-specific and overall quality of life. In this context, solving these problems is very important for the quality of care. In this regard, literature reviews on the subject have been made, and it has been observed that studies covering the entire perioperative process in patients with thyroidectomy and providing training on the problems experienced are limited and there is a significant gap regarding mobile education.It is seen that various applications have been developed in many different areas, considering that mobile-based applications will be useful in improving and maintaining health. However, no studies have been found on mobile health applications that include training to reduce patients' neck pain and discomfort levels, improve postoperative recovery, voice quality and quality of life. With the mobile-based training planned to be used in the study, it is aimed to reduce problems such as neck pain and discomfort and hoarseness experienced by patients after surgery, and to increase their recovery status and, accordingly, their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18 years or older
2. Knowing how to read and write
3. Having a planned thyroidectomy
4. Having a thyroidectomy for the first time
5. Not having a mental/visual/hearing or speech disability
6. Not having any psychiatric disease
7. Owning and using a smartphone
8. Accessing the internet at home or on the phone
9. Volunteering to participate in the study

Exclusion Criteria:

1. Not agreeing to participate in the study
2. Having a mental/visual/hearing and speech disability
3. Having a psychiatric illness
4. Having had thyroid surgery before
5. Having had complications after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2025-04-22 (Estimated); Study Completion 2025-08-22 (Estimated)

PRIMARY OUTCOMES:
Postoperative Recovery Index (ASII) | 1st day after surgery, 1st week after surgery, 4th week after surgery, 12th week after surgery
  Postoperative Healing Index Butler et al. It was developed by in 2012. ASII has five subscales. These are psychological symptoms, physical activities, general symptoms, intestinal symptoms and desire-desire symptoms. A higher score from the index indicates more difficulty in postoperative recovery, while lower scores indicate that postoperative recovery is easier.
SF-36 Quality of Life Scale | 1 day before surgery,1st day after surgery, 4th week after surgery, 12th week after surgery
  The validity and reliability study of the SF-36 Quality of Life Scale, developed by Rand Corporation in 1992 to evaluate the quality of life, in Turkish society was conducted by Pınar. SF-36; It examines the sub-dimensions of physical function, social function, physical role difficulty, emotional role difficulty, mental health, vitality/fatigue, pain, and general health perception in 36 items. Scores of the subscales range from 0 to 100, and a low score indicates poor health status. The scale is Likert type, except for some items, and there are items that include thoughts about the change in health considering the last 4 weeks. The fourth and fifth questions in the scale are evaluated with yes/no, and the other questions are evaluated with Likert type (3-point, 5-point, 6-point) rating. The score is calculated by reversing items 1, 6, 7, 8, 9a, 9d, 9e, 9h, 11b, 11d of the scale.

SECONDARY OUTCOMES:
Visual Comparison Pain Scale(GKAÖ) | 1 day before surgery,1st day after surgery, 1st week after surgery, 4th week after surgery, 12th week after surgery
  VASS is a frequently used scale in assessing pain in patients. The patient marks his/her pain on a 10 cm ruler with "no pain" written on one end and "unbearable pain" written on the other end. The use of the scale should be explained well to the patient. The patient is told that there are two extreme points on the scale and to mark the place between these points that corresponds to the severity of his pain. The distance between the beginning of "no pain" and the point marked by the patient is measured and recorded in cm.
Turkish- Computer System Usability Questionnaire Short Version (TCSUQ- SV) | 1 day before surgery, 12th week after surgery
  Turkish- Computer System Usability Questionnaire Short Version (TCSUQ-SV) was first published in 1995. Scale measures the usability of a software system; It consists of 19 items including the sub-dimensions of system usefulness, information quality and interface quality. Each item is scored as "1=strongly agree-7=strongly disagree." T-CSUQ-SV validity-reliability analyzes were conducted by US researchers Lewis and Erdinç. In the study of Erdinç and Lewis (2013), based on psychometric evaluation, the proposed short version of TCSUQ contains 13 items. For data received from groups; It can be evaluated using the average of the total score of all items, the average of the subscale scores, or the individual score average of each item.
Neck Pain and Discomfort Scale (BARÖ) | 1 day before surgery, 1st week after surgery, 4th week after surgery, 12th week after surgery
  The scale is used to evaluate pain intensity. Validity and Reliability of the Scale in Turkish Biçer et al. (2004). The scale consists of 20 items. Each item measures pain severity and evaluates the interaction of occupational, social and functional aspects of life and the presence and extent of emotional factors. Each item has a 10 cm visual analog scale. It is divided into 6 equally spaced sections with vertical bars. The score range for each item is 0-5.
Voice Handicap Index (Voice Handicap Index 10)(VHI10) | 1 day before surgery,1st day after surgery, 1st week after surgery, 4th week after surgery, 12th week after surgery
  The most well-known and widely used method in the evaluation of patients with voice problems, which is the subjective report made by the patient himself, was used by Jacobson et al. It is the Voice Handicap Index developed by . The purpose of the questionnaire is not to distinguish different pathologies from each other, but to enable the patient to evaluate his own problem. For each item, the practitioner marks a score between 0 and 4 and is rated out of a total of 40 points. As the score on the scale increases, the problems people experience with their voices increase. SHE evaluates the impact of voice disorders on patients' quality of life functionally, physiologically and emotionally. Three of the items that make up SHE-10, which is the shortened version of the Turkish Voice Handicap Index-30, are in the functional subgroup, the other three are in the physical subgroup, and four are in the emotional subgroup.

REFERENCES:
- [Background] Vrabec S, Oltmann SC, Clark N, Chen H, Sippel RS. A short-stay unit for thyroidectomy patients increases discharge efficiency. J Surg Res. 2013 Sep;184(1):204-8. doi: 10.1016/j.jss.2013.04.036. Epub 2013 May 9. PMID 23688791
- [Background] Snyder SK, Hamid KS, Roberson CR, Rai SS, Bossen AC, Luh JH, Scherer EP, Song J. Outpatient thyroidectomy is safe and reasonable: experience with more than 1,000 planned outpatient procedures. J Am Coll Surg. 2010 May;210(5):575-82, 582-4. doi: 10.1016/j.jamcollsurg.2009.12.037. PMID 20421007
- [Background] Adam MA, Thomas S, Youngwirth L, Hyslop T, Reed SD, Scheri RP, Roman SA, Sosa JA. Is There a Minimum Number of Thyroidectomies a Surgeon Should Perform to Optimize Patient Outcomes? Ann Surg. 2017 Feb;265(2):402-407. doi: 10.1097/SLA.0000000000001688. PMID 28059969
- [Background] Atasayar S, Guler Demir S. Determination of the Problems Experienced by Patients Post-Thyroidectomy. Clin Nurs Res. 2019 Jun;28(5):615-635. doi: 10.1177/1054773817729074. Epub 2017 Sep 7. PMID 28882054
- [Background] Krekeler BN, Wendt E, Macdonald C, Orne J, Francis DO, Sippel R, Connor NP. Patient-Reported Dysphagia After Thyroidectomy: A Qualitative Study. JAMA Otolaryngol Head Neck Surg. 2018 Apr 1;144(4):342-348. doi: 10.1001/jamaoto.2017.3378. PMID 29522149
- [Background] Watt T, Bjorner JB, Groenvold M, Rasmussen AK, Bonnema SJ, Hegedus L, Feldt-Rasmussen U. Establishing construct validity for the thyroid-specific patient reported outcome measure (ThyPRO): an initial examination. Qual Life Res. 2009 May;18(4):483-96. doi: 10.1007/s11136-009-9460-8. Epub 2009 Mar 14. PMID 19288224
- [Background] Takamura Y, Miyauchi A, Tomoda C, Uruno T, Ito Y, Miya A, Kobayashi K, Matsuzuka F, Amino N, Kuma K. Stretching exercises to reduce symptoms of postoperative neck discomfort after thyroid surgery: prospective randomized study. World J Surg. 2005 Jun;29(6):775-9. doi: 10.1007/s00268-005-7722-3. PMID 16078129
- See also: american thyroid association — https://www.thyroid.org/post-operative-expectations/
- See also: Nurseslabs Thyroidectomy Nursing Care Plans — https://nurseslabs.com/thyroidectomy-nursing-care-plans/